CLINICAL TRIAL: NCT02131324
Title: A Randomized, Open Label, Study to Assess the Potential for Adrenal Suppression and Systemic Drug Absorption With DFD-06 Cream Versus Clobetasol Propionate Cream, 0.05% in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: DFD06 Cream vs Clobetasol Propionate Cream, 0.05% Hypothalamic- Pituitary-Adrenal (HPA) Axis Suppression Study in Patients With Moderate to Severe Plaque Psoriasis
Acronym: HPA axis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Promius Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFD06-CD-007
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Results first posted 2018-04-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-04

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Clobetasol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clobetasol Propionate Cream, 0.05% (Active Comparator): applied twice a day for 15 days
  Interventions: Drug: Clobetasol Propionate Cream 0.05%
- DFD06 Cream (Experimental): applied twice a day for 15 days
  Interventions: Drug: DFD06 Cream

INTERVENTIONS:
Drug: DFD06 Cream
  Other Names: Clobetasol Propionate 0.025% Cream
  Arms: DFD06 Cream
Drug: Clobetasol Propionate Cream 0.05%
  Other Names: Temovate Cream
  Arms: Clobetasol Propionate Cream, 0.05%

SUMMARY:
The purpose of this study is to evaluate the potential of DFD06 cream to suppress the HPA (hypothalamic-pituitary-adrenal) axis as compared to clobetasol propionate cream, 0.05% cream when applied twice daily for 15 days.

DETAILED DESCRIPTION:
This was a 15-day, randomized, multicenter, comparator-controlled, open-label study. Approximately 50 subjects with moderate to severe plaque psoriasis were to be randomized to treatment with DFD-06 Cream or clobetasol propionate cream in a 1:1 ratio. Study products were applied twice daily for 15 days to all affected areas on the body excluding face, scalp, groin, axillae, and other intertriginous areas. Subject visits were scheduled at Screening, Baseline (Day 1), Day 8, Day 15, and Day 43 (if needed to confirm recovery). Clinical determinations of disease severity were conducted using the Investigator's Global Assessment (IGA) for overall severity at each visit.

ELIGIBILITY:
Inclusion Criteria:

Subjects must present with a clinical diagnosis of stable (at least 3 months) plaque psoriasis.

Subjects with psoriasis involving 20 to 50% Body Surface Area (BSA), not including the face, scalp, groin, axillae and other intertriginous areas.

Subjects must have an IGA grade of at least 3 (moderate) at the Baseline Visit Subjects whose results from the screening Adrenocorticotropic hormone (ACTH) stimulation test are considered normal (cortisol level >18 ug/dL at 30 minutes post stimulation) and show no other signs of abnormal HPA function or adrenal response

Exclusion Criteria:

Current diagnosis of unstable forms of psoriasis including guttate, erythrodermic, exfoliative or pustular psoriasis.

History of organ transplant requiring immunosuppression, HIV, or other immunocompromised state.

Have received treatment for any type of cancer within 5 years of the Baseline Visit except skin cancer and cervical cancer (in situ) are allowed if at least 1 year before the Baseline Visit.

Use within 60 days prior to the baseline Visit of: 1) immunosuppressive drugs (e.g., tacrolimus, pimecrolimus), or 2) systemic antipsoriatic treatment (e.g., methotrexate, cyclosporine, hydroxyurea) Use within 30 days prior to the Baseline Visit of: 1) topical antipsoriatic drugs (salicylic acid, anthralin, coal tar, calcipotriene), 2) psoralen and ultraviolet A (PUVA) therapy, 3) systemic anti-inflammatory agents (e.g., mycophenolate mofetil, sulfasalazine, 6-thioguanine), or 4) ultraviolet B (UVB) therapy.

Use within 30 days prior to the Screening Visit of any product containing corticosteroids. Inhaled, intraocular, intranasal, etc. steroids are not allowed.

Subjects who have an abnormal sleep schedule or work at night. Subjects with a known history of acute adrenal crisis, Addison's disease or decreased adrenal output, low pituitary function or pituitary tumors.

Subjects who have a history of an adverse reaction to cosyntropin injection or similar test reagents.

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05-08 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Sidgiddi, MD, Study Director — Dr. Reddy's Laboratories, Inc
Locations (15):
- United States (15):
  - Advanced Research Associates, Glendale, Arizona
  - Agave Clinical Research, LLC, Mesa, Arizona
  - T. Joseph Raoof, MD, Inc., Encino, California
  - International Dermatology Research, Inc., Miami, Florida
  - FXM Research Corp., Miami, Florida
  - FXM Research Miramar, Miramar, Florida
  - Belleair Research, Pinellas Park, Florida
  - Forward Clinical Trials, Tampa, Florida
  - Marietta Dermatology Clinical Research, Inc., Marietta, Georgia
  - Determatology Specialists Research, LLC, Louisville, Kentucky
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Dermatology Consulting Services, High Point, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Radiant Research, Inc., Greer, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Washout was needed at Screening Visit if prohibited therapies were in use.
  The screening adrenocorticotropic hormone (ACTH) stimulation test was conducted at least 14 days and no more than 28 days prior to the Baseline Visit.
Groups:
- Comp01: applied twice a day for 15 days
  Comp01
- DFD06 Cream: applied twice a day for 15 days
  DFD06 Cream
Period: Overall Study
Arm/Group | Comp01 | DFD06 Cream
Started | 24 (2 subjects randomized into Comp01 not included in analysis as there was no post-baseline information) | 26 (2 subjects randomized into DFD-06 not included in analysis as there was no post-baseline information)
Analyzed | 22 | 24
Completed | 22 | 23
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- DFD06: DFD06 Active
- Comp01: Comp01 Comparator
- Total: Total of all reporting groups
Arm/Group | DFD06 | Comp01 | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 22 | 45
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (14.5) | 50.9 (11.2) | 47.0 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 17 | 14 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 13 | 27
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 24 | 22 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 22 | 46
Body Surface Area (BSA) affected by psoriasis [Mean (Standard Deviation); unit: cm^2] — Population: Two subjects dropped out of the study in each arm.
  cm^2 | 26.5 (8.6) | 27.0 (8.3) | 26.8 (8.4)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects With HPA Axis Suppression.
Description: HPA axis suppression as measured by serum cortisol levels post cosyntropin test (ACTH test)
Time Frame: Day 15
Population: All summaries and analyses were performed on the safety population. All subjects who received at least one confirmed dose of study product and provided any post-baseline safety information were included in the safety population. No imputation was made for missing safety data.
Measure: Number; unit: percentage of participants
Groups:
- Clobetasol Propionate Cream, 0.05%: applied twice a day for 15 days
  Clobetasol Propionate Cream, 0.05%
Arm/Group | Clobetasol Propionate Cream, 0.05% | DFD06 Cream
Number analyzed (Participants) | 22 | 24
percentage of participants | 36.4 | 12.5
Statistical Analysis 1: Comparison: Clobetasol Propionate Cream, 0.05% vs DFD06 Cream; Two-sided hypothesis testing was conducted for all the tests. Resulting p-values less than 0.05 were considered statistically significant unless noted otherwise. No adjustments of p values were made for multiple comparisons; Test type: Equivalence — Two-sided hypothesis testing was conducted for all the tests. Resulting p-values less than 0.05 were considered statistically significant unless noted otherwise. No adjustments of p values were made for multiple comparisons; p = 0.086, ANOVA

ADVERSE EVENTS:
Groups:
- Clobetasol Propionate Cream, 0.05%: applied twice a day for 15 days
  Clobetasol Propionate Cream 0.05%
Arm/Group | Clobetasol Propionate Cream, 0.05% | DFD06 Cream
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/24
Other Adverse Events (participants affected / at risk) | 11/22 | 5/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clobetasol Propionate Cream, 0.05% (N=22) | DFD06 Cream (N=24)
Injury/Stab Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Stab wound at right lower quadrant of abdomen
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clobetasol Propionate Cream, 0.05% (N=22) | DFD06 Cream (N=24)
HPA axis suppression (Endocrine disorders) | 8 (8) | 3 (3)
Application site pain (General disorders) | 2 (2) | 0 (0)
Application site pruritus (General disorders) | 1 (1) | 0 (0)
Dehydroepiandrosterone sulfate dicreased (Investigations) | 6 (6) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less